CLINICAL TRIAL: NCT07382687
Title: A Phase 3, Multicenter, Randomized, Open-label, Active-controlled Trial of Famitinib Combined With SHR-A1811, Versus SHR-A1811 for CDK4/6 Inhibitors-resistent Advanced HR+/HER2- Breast Cancer With SNF4 Subtype
Brief Title: Famitinib Combined With SHR-A1811, Versus SHR-A1811 for CDK4/6 Inhibitors-resistent Advanced HR+/HER2- Breast Cancer With SNF4 Subtype
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Zhimin Shao, Director of General Surgery of Fudan Shanghai Cancer Center, Fudan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SCHBCC-N099; MA-BC-III-133 (Other: Breast cancer institute of Fudan University Cancer Hospital)
Record Dates: First submitted 2026-01-27; First posted 2026-02-03 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Active Comparator): SHR-A1811
  Interventions: Drug: SHR-A1811
- Experimental (Experimental): Famitinib+SHR-A1811
  Interventions: Drug: Famitinib+SHR-A1811

INTERVENTIONS:
Drug: SHR-A1811 — SHR-A1811 4.8mg/kg iv q3w
  Arms: Control
Drug: Famitinib+SHR-A1811 — Famitinib 10mg po qd SHR-A1811 4.8mg/kg iv q3w
  Arms: Experimental

SUMMARY:
This study is a prospective, open-label, multicenter, randomized controlled Phase III clinical trial. This study aims to investigate the efficacy and safety of Famitinib combination with SHR-A1811 in CDK4/6 inhibitors-resistent advanced HR+/HER2- breast cancer with SNF4 subtype.

ELIGIBILITY:
Inclusion Criteria:

1. Women aged 18-70 years old;
2. Histologically confirmed HR+/HER2- invasive breast cancer (specific definition: ER >10% of tumor cells positive by immunohistochemistry is defined as ER positive, PR >10% of tumor cells positive by immunohistochemistry is defined as PR positive, ER and/or PR positive is defined as HR positive; HER2 low expression or ultra-low expression [FISH/CISH- and IHC+/++ or IHC 0 but with ≤10% of tumor cells showing incomplete and weak cell membrane staining]);
3. SNF4 subtype definition: SNF4 subtype confirmed by digital pathology of H&E sections and artificial intelligence;
4. Locally advanced breast cancer (unresectable locally) or recurrent and metastatic breast cancer;
5. Have used CDK4/6 inhibitors in the recurrent and metastatic stage, or have relapsed and metastasized within 1 year of adjuvant CDK4/6 inhibitor use;
6. At least one measurable lesion according to RECIST 1.1 criteria (≥20 mm by conventional CT scan, ≥10 mm by spiral CT scan, and the measurable lesion has not received radiotherapy), or in the absence of measurable lesions, have non-measurable osteolytic or mixed (osteolytic + osteoblastic) bone lesions;
7. Basic normal major organ function, meeting the following conditions: (a) Blood routine examination standards need to meet: HB ≥90 g/L (no blood transfusion within 14 days); ANC ≥1.5×109/L; PLT ≥75×109/L;(b) Biochemical examination needs to meet the following standards: TBIL ≤1.5×ULN (upper limit of normal value); ALT and AST ≤3×ULN; if there is liver metastasis, ALT and AST ≤5×ULN; serum Cr ≤1.5×ULN, endogenous creatinine clearance rate >50 ml/min (Cockcroft-Gault formula);(c) Electrocardiogram: Fridericia's corrected QT interval (QTcF) < 450 ms for men and < 470 ms for women;
8. ECOG score ≤2, and expected survival ≥3 months;
9. Female subjects who are capable of bearing children need to adopt a medically approved contraceptive measure during the study treatment period and for at least 3 months after the last use of study medication;
10. Subjects voluntarily join this study, sign the informed consent form, have good compliance and cooperate with follow-up

Exclusion Criteria:

1. Uncontrolled central nervous system metastasis (referring to symptoms or the need for corticosteroids or mannitol to control symptoms);
2. Left ventricular ejection fraction (LVEF) <50% (as determined by echocardiography);
3. History of any of the following cardiac diseases: (1) angina pectoris; (2) clinically significant arrhythmia requiring medication; (3) myocardial infarction; (4) heart failure; (5) any other cardiac disease deemed unsuitable for participation in this trial by the investigator;
4. previously suffered from clinically significant pulmonary diseases, including but not limited to interstitial pneumonia, pneumonia, pulmonary fibrosis, and radiation pneumonia (excluding radiation changes that do not require corrective treatment), or have been found to have suspected such diseases during screening period examinations;
5. Individuals who have received radiotherapy, chemotherapy, surgical treatment (excluding minor outpatient surgeries such as placement of vascular access) or other targeted and immunotherapy treatments for advanced HR+/HER2- breast cancer within 3 weeks prior to the first administration of study drugs;
6. Individuals who have ongoing ≥ Grade 1 adverse reactions due to previous treatments. Exceptions to this include hair loss or conditions that the investigator deems should not be excluded. Such cases should be clearly documented in the investigator's notes;
7. Pregnant or lactating patients;
8. Individuals who have had malignant tumors within the past three years (excluding cured basal cell carcinoma of the skin and carcinoma in situ of the cervix);
9. Significant comorbidities, including mental illnesses that the investigator believes may adversely affect the patient's participation in the study;
10. Patients with a history of gastrointestinal bleeding within the past 6 months or a clear tendency for gastrointestinal bleeding, such as esophageal varices with bleeding risk, localized active ulcer lesions, and occult blood in stool ≥ (++), are not eligible for enrollment; if occult blood in stool is (+), gastroscopy is required;
11. Patients who have experienced abdominal fistula, gastrointestinal perforation, or abdominal abscess within 28 days before participating in this study;
12. Patients with imaging findings indicating tumor invasion around important blood vessels or, in the judgment of the investigator, a high likelihood of tumor invasion during treatment causing fatal massive hemorrhage;
13. Patients who have experienced arterial/venous thromboembolic events within one year before screening, such as cerebrovascular accidents (including transient ischemic attacks), deep venous thrombosis (excluding cases where venous thrombosis caused by venous catheterization during previous chemotherapy has been judged by the investigator to have healed), and pulmonary embolism;
14. Patients with urine routine test showing urine protein ≥++ or confirmed 24-hour urine protein quantitation >1.0g;
15. Patients with hypertension who cannot be brought to normal range by antihypertensive medication (systolic blood pressure >140mmHg, diastolic blood pressure >90mmHg);
16. Patients with swallowing difficulties, chronic diarrhea, and intestinal obstruction, which affect drug administration and absorption in various ways;
17. Patients with third-space effusion that cannot be controlled by drainage or other methods (such as large amounts of pleural effusion and ascites);
18. Patients with allergic constitution, or known history of allergy to components of the study drugs; or patients allergic to other monoclonal antibodies;
19. Patients with known active HBV or HCV infection or HBV DNA ≥500, or chronic phase with abnormal liver function;
20. Any other situations where the investigator deems the patient unsuitable for participation in this study.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 248 (Estimated)
Dates: Start 2026-02-26 (Estimated); Primary Completion 2028-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival(PFS) Based on Investigator Assessment | From the date of randomization to the earliest date of the first objective documentation of radiographic disease progression or death due to any cause, up to approximately 3 years

SECONDARY OUTCOMES:
Overall survival (OS) | From the date of randomization up to the date of death due to any cause, up to approximately 3 years
Objective response rate (ORR) | From screening and every 6 weeks up to withdrawal of subject consent, progressive disease (PD), or unacceptable toxicity, up to approximately 3 years
Clinical benefit rate(CBR) | From screening and every 6 weeks up to withdrawal of subject consent, progressive disease (PD), or unacceptable toxicity, up to approximately 3 years
Duration of Response(DOR) | From the date of the first documented objective response (CR or PR) to the first documented disease progression or death, whichever occurs first, up to approximately 3 years
Time to Response(TTR) | from randomization to the achievement of first objective response, up to approximately 3 years
Treatment-Emergent Adverse Events (TEAEs) and Treatment-Emergent Serious Adverse Events(TESAEs) | From first dose of study drug (Day 1) up to approximately 3 years

CONTACTS AND LOCATIONS:
Locations (1):
- Breast cancer institute of Fudan University Cancer Hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: Undecided